CLINICAL TRIAL: NCT04275778
Title: Evaluation of the Benefit of Adjuvant Treatment With Hydroxychloroquine to the Usual Medical Management for Obtaining an Uncomplicated Term Pregnancy in Primary Obstetric Antiphospholipid Syndrome
Brief Title: HYDROxychloroquine in Syndrome Primary AntiPhospholipid
Acronym: HYDROSAPL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160944J
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Antiphospholipid Syndrome in Pregnancy; Anticoagulants
Keywords: APS; Anticoagulants; Pregancy; Heparin Low-Molecular-Weight; Aspirin
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Group 1 : Hydroxychloroquine Group 2 : Placebo d'hydroxychloroquine Hydroxychloroquine or placebo will be performed at 2 pills (400 mg) per day, during the pregnancy, and stopped at delivery.
  The conventional treatment will be the same in the 2 groups:
  * aspirin 100 mg/day will begin , the preference at the preconception, and continued during pregnancy and will be stopped at 35 weeks of gestation.
  LMWH enoxaparin 4000 UI/day will begin as soon as possible after confirmation of the pregnancy, and will be continued during 6 weeks postpartum.
Who Masked: Participant, Investigator
Masking Description: Hydroxychloroquine and placebo will be provided by "AGEPS" which outsources these drugs fabrication. The "AGEPS" outsources operations which are technically non-feasible locally, or if the volume or logistical constraints are inconsistent with the balance of its human and material resources.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine will be prescribed upon confirmation of pregancy at a dosage of 400 mg / day. Either in 2 doses (1 tablet of 200 mg in the morning and 1 tablet of 200 mg in the evening). Or in a single take: 2 tablets of 200 mg.
  Treatment will be continueted during the pregnancy and will be stopped at delivery.
  Interventions: Drug: Plaquenil 200Mg Tablet
- Placebo group (Placebo Comparator): Placebo will be prescribed upon confirmation of pregancy at a dosage of 400 mg / day. Either in 2 doses (1 tablet of 200 mg in the morning and 1 tablet of 200 mg in the evening). Or in a single take: 2 tablets of 200 mg.
  Treatment will be continueted during the pregnancy and will be stopped at delivery.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Plaquenil 200Mg Tablet — Hydroxychloroquine will be taken at a dosage of 400 mg / day until delivery
  Arms: Hydroxychloroquine
Drug: Placebo oral tablet — placebo will be taken at a dosage of 400 mg / day until delivery
  Arms: Placebo group

SUMMARY:
Antiphospholipid syndrome (APS) is defined by thrombosis or obstetric complication (≥ 3 spontaneous miscarriages or fetal death or prematurity <34 weeks gestation-related amenorrhea (SA)) associated with antiphospholipid antibodies. The rate of term pregnancies has been improved by conventional treatment (aspirin 100 mg / day with low molecular weight heparin (LMWH) in an isocoagulant dose) to almost 75%. In the PROMISSE study, when considering progressive pregnancies after 20 weeks, 19% of pregnancies presented at least one complication despite the treatment (maternal, fetal or neonatal complications) related to APS. In the European APS register, maternal complications and IUGR were observed in 13% of cases, and prematurity in approximately 14% of cases despite treatment. In a previous study of 72 pregnancies during a LAS, we observed, under aspirin and LMWH, 25% of fetal losses, and 10% of at least one maternal and / or fetal complication or prematurity. The presence of lupus, a history of thrombosis, a circulating anticoagulant (ACC) and a triple positivity of antiphospholipids are considered to be factors associated with a poor obstetrical prognosis. Hydroxychloroquine (HCQ) has anti-inflammatory and anti-thrombotic properties. In vitro studies have shown that HCQ is able to restore the expression of placental annexin V, which has an anticoagulant effect and prevent the attachment of antiphospholipid antibodies to the placenta.

HCQ during lupus decreases the thrombotic risk and its usefulness during thrombotic APS has been shown in a French series. In a European study, the addition of the HCQ to conventional treatment improved term pregnancies by 70% in the event of refractory APS. Its use during pregnancies of patients with lupus, the numerous data on tolerance during pregnancy and the follow-up of children born to mothers exposed to the HCQ demonstrates a reassuring tolerance profile for the mother and the fetus.

The objective of this clinical trial is to evaluate the benefit of addition or no of hydroxychloroquine to conventional treatment in obstetric APS.

DETAILED DESCRIPTION:
The consecutive patientes with APS will be recruited in different ways based on daily practice; Patients fulfilling all criteria may be randomized following receipt of written informed consent.

The randomization will be stratified by center and by, the presence of anticoagulant antibody.

Te included patients will be randomized to receive conventional APS treatment (aspirin with low-molecular-weight heparin) combined with hydroxychloroquine or placebo.

In the two groups, the hydroxychloroquine or placebo will be initiated in the patients with ongoing pregnancy (≤14 week of gestation).

After the inclusion visit, the patients will be followed by the investigator every months until the end of the pregnancy and at 6 weeks postpartum.

At each visit, a clinical examination, routine biological analysis, APL antibody and complement determination will be performed. Hydroxychloroquine blood levels, PFA, Xa inhibition,and treatment adherence will be assessed during pregnancy.

At Inclusion :

- Maternal blood samples 20 ml of blood will be collected at the same time as the sample routinely collected just before delivery when the women are perfused.

At delivery

- Cord fluid : will be collected at the same as cord fluid pH is routinely measured just after delivery. The aliquots previously labelled and stowed in the specific boxes for the study will be stored locally and will be transported to the "Centre de Ressources Biologiques"(CRB) of the Saint Antoine Hospital. Last visit for children : At 12 months The patient will be contacted by phone by the local medical team to collect the following data: Children's anthropometric data; safety data ; possible hospitalization..

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Spontaneous consecutive pregnancy ongoing before the 14th week of gestation

  -- SAPL obstetrics (modified Sapporo criteria = Sydney criteria) with fetal death ≥10 weeks of gestation without further explanation; and / or preeclampsia (or HELLP syndrome) and / or prematurity <34SA with placental insufficiency (with or without thrombotic SAPL)
* Signed informed consent

Exclusion Criteria:

* Other SAPL subgroups: early isolated miscarriages <10 weeks
* Contraindication to hydroxychloroquine:

  * retinopathy,
  * hypersensitivity to chloroquine or hydroxychloroquine or to any of the other ingredients especially lactose
* Associated systemic lupus, associated Sjogren syndrome
* Treatment with hydroxychloroquine in progress
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Lack of Social Insurance

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2024-10-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of term pregnancies with a eutrophic child | at delivery
  eutrophic child = a full term birth without maternal, fetal or neonatal complications

CONTACTS AND LOCATIONS:
Overall Officials: Arsène MEKINIAN, MD, Principal Investigator — Internal Medecine_Hospital Saint Antoine
Locations (1):
- Hopital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Irastorza G, Crowther M, Branch W, Khamashta MA. Antiphospholipid syndrome. Lancet. 2010 Oct 30;376(9751):1498-509. doi: 10.1016/S0140-6736(10)60709-X. Epub 2010 Sep 6. PMID 20822807
- [Background] Fain O, Mekinian A. [Antiphospholipid syndrome]. Rev Prat. 2011 Nov;61(9):1261-2. No abstract available. French. PMID 22308813
- [Background] Mekinian A, Lachassinne E, Nicaise-Roland P, Carbillon L, Motta M, Vicaut E, Boinot C, Avcin T, Letoumelin P, De Carolis S, Rovere-Querini P, Lambert M, Derenne S, Pourrat O, Stirnemann J, Chollet-Martin S, Biasini-Rebaioli C, Rovelli R, Lojacono A, Ambrozic A, Botta A, Benbara A, Pierre F, Allegri F, Nuzzo M, Hatron PY, Tincani A, Fain O, Aurousseau MH, Boffa MC. European registry of babies born to mothers with antiphospholipid syndrome. Ann Rheum Dis. 2013 Feb;72(2):217-22. doi: 10.1136/annrheumdis-2011-201167. Epub 2012 May 15. PMID 22589374
- [Background] Mekinian A, Loire-Berson P, Nicaise-Roland P, Lachassinne E, Stirnemann J, Boffa MC, Chollet-Martin S, Carbillon L, Fain O. Outcomes and treatment of obstetrical antiphospholipid syndrome in women with low antiphospholipid antibody levels. J Reprod Immunol. 2012 Jun;94(2):222-6. doi: 10.1016/j.jri.2012.02.004. Epub 2012 Mar 3. PMID 22386067
- [Background] Mekinian A, Lazzaroni MG, Kuzenko A, Alijotas-Reig J, Ruffatti A, Levy P, Canti V, Bremme K, Bezanahary H, Bertero T, Dhote R, Maurier F, Andreoli L, Benbara A, Tigazin A, Carbillon L, Nicaise-Roland P, Tincani A, Fain O; SNFMI and the European Forum on Antiphospholipid Antibodies. The efficacy of hydroxychloroquine for obstetrical outcome in anti-phospholipid syndrome: Data from a European multicenter retrospective study. Autoimmun Rev. 2015 Jun;14(6):498-502. doi: 10.1016/j.autrev.2015.01.012. Epub 2015 Jan 21. PMID 25617818